CLINICAL TRIAL: NCT06410014
Title: Assessment of Overall Functioning in Patients With Complex Health Issues
Acronym: CPH-Func
Status: Recruiting | Type: Observational
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Principal Investigator, Anna Karnøe Knudsen, Prinicipal Investigator, University Hospital Bispebjerg and Frederiksberg
Other Study IDs: H23030964
Record Dates: First submitted 2024-03-11; First posted 2024-05-10 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Activities of Daily Living; Surveys and Questionnaires; ADL Motor Skills; Disability Evaluation; Health Status; Muscle Strength; Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participating patients: All patient who have consented to participate in the study
  Interventions: Other: No intervention is performed

INTERVENTIONS:
Other: No intervention is performed — The study is observational

SUMMARY:
The overall aim of the study is to assess whether each outcome measures the same aspect of overall functioning or contributes with different aspects. More specifically, the aim of this study is to investigate the correlation between each single instrument.

During study period all patients presenting at our clinic will be offered to participate in the study. Patients will be included in the study when referred to the department of Social Medicine and providing written informed consent to participate in the study. Inclusion will continue until 100 patients have completed an AMPS test. All participants will, apart from standard procedure, be asked to complete:

* An AMPS-test
* ADL-Q (Questionnaire concerning Activities of Daily Living)
* ADL-I (Interview based questionnaire concerning Activites of Daily Living)

As standard procedure all participants will also perform/complete:

* 30 seconds chair stand test (30sCST)
* Hand grip strength (HGS)
* Evaluation of ambulation (Cumulated Ambulation Score /CAS)
* WORQ (Work Rehabilitation Questionnaire)

To obtain the aim of the study correlation-analysis will be performed to investigate the relationship between each included instruments.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred by a municipality to the Department of Social Medicine at Bispebjerg and Frederiksberg Hospital for a clinical assessment (Klinisk Funktion) who provide written consent to participate.

Exclusion Criteria:

* Insufficient ability to communicate either in written or oral Danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The department of social medicine receives patients referred by the municipality for a general clinical examination and an assessment of overall functioning (Klinisk Funktion). The criteria of referral are a need of a medical assessment of complex health issues and the impact on functioning and/or symptoms with no equivalent objective findings. Generally, the patients referred are characterized by complex health issues and several years of unemployment. The conclusion, which consists of a medical review and an assessment of overall functioning, is sent to the municipality and used e.g., in their assessment of workability and social insurance.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of Motor and Process Skills (AMPS) | Within 21 days from baseline
  Based on observation of 2 ADL tasks the quality of 16 motor and 20 process skills are scored on a four-point ordinal scale. Using Rasch analysis the raw ordinal scores are converted into two overall ADL ability measures, representing ADL motor and ADL process ability expressed in logits.

SECONDARY OUTCOMES:
30 seconds chair stand test | Baseline
  Total number of stands performed in 30 seconds
Hand Grip strength | Baseline
  Measured in kilograms
Cumulated Ambulation Score (CAS) | Baseline
  Scoring of three mobility activities on a three point ordinal scale (zero to 2). The scores are summed resulting in a total score ranging from 0 to 6.
ADL-I | Within 21 days from baseline
  Raw data collected in the interview is scored on a four-point ordinal scale and subsequently converted into a linear measure of self-reported ADL ability expressed in logits (log-odds probability units).
ADL-Q | Within 21 days from baseline
  Raw data collected in the questionnaire is scored on a four-point ordinal scale and subsequently converted into a linear measure of self-reported ADL ability expressed in logits (log-odds probability units).
Work Rehabilitation Questionnaire (WORQ) | The questionnaire is responded one time during a periode ranging from 7 days prior to baseline until 21 days after baseline
  The questionnaire consists of 17 items on sociodemographic topics and 40 items related to overall functioning. The 40 items are each scored on a response scale ranging from 0 to 10. The results are summed in four linear subscales addressing emotion, cognition, dexterity and mobility. A total sum score is performed.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Renneberg, DMSc, Study Chair — Department of Social Medicine; Anna Karnøe Knudsen, M.D., Principal Investigator — Department of Social Medicine
Locations (1):
- Afdeling for Socialmedicin, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2024-03-11): https://cdn.clinicaltrials.gov/large-docs/14/NCT06410014/Prot_000.pdf